CLINICAL TRIAL: NCT00561561
Title: Sensorimotor Gating in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Erica Duncan, MD, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00021861
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Prepulse Inhibition; Acoustic Startle
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Subjects with schizophrenia
  Interventions: Behavioral: Acoustic startle testing
- 2 (Active Comparator): Health controls
  Interventions: Behavioral: Acoustic startle testing
- 3 (Active Comparator): Family members of subjects with schizophrenia
  Interventions: Behavioral: Acoustic startle testing
- 4 (Active Comparator): Family members of healthy controls
  Interventions: Behavioral: Acoustic startle testing

INTERVENTIONS:
Behavioral: Acoustic startle testing — recording of eyeblink component of acoustic startle reflex with small surface electrodes during presentation of acoustic stimuli through headphones

SUMMARY:
This study is looking at problems people sometimes have taking in information from their senses. Specifically, we are comparing the way in which people diagnosed with schizophrenia process sound information, compared with people who have never been diagnosed with a psychiatric disorder. When people hear a loud sound they sometimes feel startled, and when they feel startled they usually blink their eyes. However, if they hear a softer sound shortly before the loud one they may not blink their eyes - in other words, the eye-blink response is smaller. When this happens it's called prepulse inhibition of startle. In this study, we want to measure the startle response and prepulse inhibition of startle in individuals diagnosed with schizophrenia versus individuals not diagnosed with schizophrenia. We also want to find out whether people show the same amount of prepulse inhibition of startle as other members of their family.

DETAILED DESCRIPTION:
Patients with schizophrenia have difficulty screening out irrelevant stimuli, and often have the experience of sensory flooding. These "gating deficits" may contribute to the thought disorder, cognitive fragmentation and hallucinations which are so debilitating to these individuals. The acoustic startle response is a reflex contraction of the skeletal muscles in response to a sudden acoustic stimulus. It occurs across mammalian species and can be easily measured. The modulation of this reflex by a preliminary nonstartling stimulus is termed prepulse inhibition of acoustic startle (PPI), a paradigm which is used as an operational measure of sensorimotor gating. In consonance with the schizophrenia symptoms that are suggestive of gating deficits, many patients with schizophrenia have deficits in PPI when compared to healthy controls. The brain regions that modulate PPI include the hippocampus and prefrontal cortex, areas that are implicated as being abnormal in schizophrenia. Our prior work and work from other labs suggests that PPI impairment in schizophrenia does not improve with treatment and hence may be a trait related abnormality. Work from our current funding period supports our original hypothesis, namely that impaired PPI exhibits familial association. Specifically, we are finding that PPI in first degree family members of subjects with schizophrenia is impaired. Further work is needed in order to establish that PPI impairment is heritable.

An endophenotype is a measurable trait or phenotype detectable by a biological test. Using an endophenotype rather than presence or absence of disease is a powerful tool in the study of diseases with complex polygenic etiologies such as schizophrenia. Progress in the genetics of schizophrenia is greatly confounded by the difficulty in identifying individuals who carry genes contributing to schizophrenia. Incomplete penetrance and the fact that both heritable and environmental factors interact to produce the disease add to this difficulty. This means that some individuals carrying vulnerability genes for schizophrenia who fail to exhibit robust symptoms will be classified erroneously as unaffected in genetic studies, confounding attempts to reliably define the heritable phenotype. The phenomenon of incomplete penetrance is exhibited by the finding that the risk of schizophrenia is the same for children of affected and nonaffected monozygotic twins. The polygenic etiology of schizophrenia makes it unlikely that a pooled sample of individuals defined by the presence of schizophrenia will greatly overlap in the vulnerability genes that they carry. The goal of the endophenotype approach is to narrow the defined phenotype so that a more homogeneous genotype is expected, making it much more fruitful and to conduct genetic studies.

We hypothesize that impaired PPI will prove to be a heritable endophenotype in schizophrenia. Based on our work accomplished during the current funding period, we now propose to further develop this line of research by conducting a heritability analysis of PPI. Our field is greatly in need of this work as a prelude to endophenotype-based genetic studies. We will accomplish our important goal by collecting and characterizing a cohort of healthy controls and their families, and by expanding our sample of schizophrenia subjects and their families. We will collect diagnostic, symptom, cognitive, pedigree, and PPI data all subjects, and will collect blood and extract DNA for future genetic analyses. We will use a family based strategy to investigate the pattern and degree of heritability of impaired PPI in families of schizophrenia and control probands.

This project will provide the necessary next step in advancing the use of impaired PPI as a powerful tool for the discovery of vulnerability genes contributing to schizophrenia. Currently available treatments for this devastating disorder are sadly inadequate. Our medications are virtually ineffective for a subset of our patients. The discovery of vulnerability genes and of a method for biological subtyping of patients will allow our field to develop genetically informed new treatments that specifically target particular subtypes of patients. This approach is our best hope for bringing relief to patients suffering from this disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a Schizophrenia Spectrum disorder OR no history of Psychiatric Illness

Exclusion Criteria:

* History of head injury with loss of consciousness of more than 5 minutes
* History of neurological disease (ex. meningitis, encephalitis)
* Drug or alcohol abuse within the last 3 months
* Hearing loss
* Non-correctable vision problems
* Current cancer treatment (radiation or chemotherapy currently ongoing)
* History of Post Traumatic Stress Disorder
* Diagnosis of HIV or AIDS
* Uncontrolled diabetes
* History of seizures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2001-06; Primary Completion 2011-08-26 (Actual); Study Completion 2011-08-26 (Actual)

PRIMARY OUTCOMES:
Prepulse inhibition of acoustic startle | Day 1 Post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Erica Duncan, MD, Principal Investigator — Atlanta VA Medical Center, Emory University Dept of Psychiatry & Behavioral Sciences
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No